CLINICAL TRIAL: NCT04645511
Title: A Placebo Controlled Randomised Study of the Balloon Sinuplasty Efficiency in Chronic or Recurrent Maxillary Rhinosinusitis.
Brief Title: Balloon Sinuplasty Efficiency in Maxillary Rhinosinusitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R20026
Record Dates: First submitted 2020-06-26; First posted 2020-11-27 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-05

CONDITIONS: Maxillary Sinusitis; Sinusitis, Chronic; Sinusitis Recurrent; Eustachian Tube Dysfunction
Keywords: Balloon sinuplasty
MeSH Terms: conditions — Maxillary Sinusitis; Sinusitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, placebo-controlled, double-blinded clinical study
Who Masked: Participant, Investigator
Masking Description: Throughout the study, both the patients and the examining doctors are blinded regarding the patients' group status. The patients are randomized using a MINIM-program by a person, who doesn't participate in treating or following up the patients. The operating doctor only operates the patients but doesn't participate in the pre- or postoperative evaluation. The information, whether the patient had a placebo procedure or the balloon sinuplasty procedure, is not written in the patient's medical record but only on the Surgery form and the form is sealed in an envelope. The envelope is only opened in the end of the 12-month follow-up period. The patient's eyes are covered with moist gauze dressing pads during the operation and the staff pays extreme attention not to let the patient know his/her group status. Neither do the examining doctors know the patient's group status during the 12 month follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chronic sinusitis: Balloon sinuplasty (Experimental): 30 patients with chronic maxillary sinusitis that are randomized to be treated with the real Balloon sinuplasty procedure of maxillary sinuses.
  Interventions: Procedure: Balloon sinuplasty of maxillary sinuses
- Chronic sinusitis: Placebo (Sham Comparator): 30 patients with chronic maxillary sinusitis that are randomized to be treated with sham surgery.
  Interventions: Procedure: Sham surgery
- Recurrent sinusitis: Balloon sinuplasty (Experimental): 30 patients with recurrent maxillary sinusitis that are randomized to be treated with the real Balloon sinuplasty procedure of maxillary sinuses.
  Interventions: Procedure: Balloon sinuplasty of maxillary sinuses
- Recurrent sinusitis: Placebo (Sham Comparator): 30 patients with recurrent maxillary sinusitis that are randomized to be treated with sham surgery.
  Interventions: Procedure: Sham surgery

INTERVENTIONS:
Procedure: Balloon sinuplasty of maxillary sinuses — A shapeable tip of the balloon dilatation device (Entellus XprESS LoProfile; Stryker Corporation, Kalamazoo, Michigan, U.S.A.), with maxillary bending, is inserted into the maxillary sinus ostium. Then guided with the tip, a flexible balloon (6 mm x 20 mm) is gently inserted into the ostium and inflated up to 12 atm for 15 seconds. The dilatation is repeated one more time. The same procedure is performed for both maxillary sinuses.
  Arms: Chronic sinusitis: Balloon sinuplasty; Recurrent sinusitis: Balloon sinuplasty
Procedure: Sham surgery — The middle meatus is gently palpated with a curved suction tip (the tip is not connected to a suction unit). The curved suction tip is placed medial to the uncinate process. In order to create a better placebo effect, the operating doctor says: "Now inflate the balloon up to 12 atm for 15 seconds." After 15 seconds the doctor says: "Deflate the balloon." This is repeated one more time. Similar procedure is carried out on both sides.
  Arms: Chronic sinusitis: Placebo; Recurrent sinusitis: Placebo

SUMMARY:
This study is a prospective, randomized, placebo-controlled, double-blinded clinical study. The balloon sinuplasty treatment is compared to placebo effect in chronic or recurrent maxillary sinusitis. The purpose is to find out the efficacy of balloon sinuplasty of maxillary sinuses and the patients who get the best benefit from balloon sinuplasty. The investigators also want to find out if balloon sinuplasty of maxillary sinuses improves Eustachian tube dysfunction. The study is executed in the Department of Ear and Oral Diseases, Tampere University Hospital. 120 patients who have either recurrent acute or chronic rhinosinusitis without nasal polyposis and whose sinusitis is limited mainly into maxillary sinuses, are recruited in the study. The patients are allocated either into the chronic maxillary sinusitis (60 patients) or the recurrent maxillary sinusitis (60 patients) branch of the study. Then, the patients are consecutively randomized into two treatment groups in the proportion of 1 to 1: A) Balloon sinuplasty group and B) Placebo group. The treatment is performed according to the patient's group status and all the patients are followed 12 months postoperatively.

The effect of balloon sinuplasty treatment in chronic maxillary rhinosinusitis is going to be measured primarily with the Sino-Nasal Outcome Test (SNOT-22). In recurrent acute maxillary rhinosinusitis, the effect of balloon sinuplasty treatment will be measured primarily with the number of acute rhinosinusitis infections. Besides this, number of antibiotic treatments and sick leaves are inquired, Visual Analog Scale (VAS) and Eustachian Tube Dysfunction Questionnaire (ETDQ-7) are used, rhinomanometry, Cone Beam Computed Tomography (CBCT), tympanometry, tubomanometry, nasal endoscopy and general evaluation of the patients clinical ORL-status are performed. Also pre- and postoperative biopsies are taken from the middle turbinates.

DETAILED DESCRIPTION:
This study is a prospective, randomized, placebo-controlled, double-blinded clinical study. The purpose of the study is to compare the balloon sinuplasty treatment to placebo effect in chronic or recurrent maxillary sinusitis and to find out the efficacy of balloon sinuplasty in different stages of rhinosinusitis (recurrent vs. chronic). The goal is to find out the patients who get the best benefit from balloon sinuplasty. The investigators also want to find out if balloon sinuplasty of maxillary sinuses improves Eustachian tube dysfunction.

The study is executed in the Department of Ear and Oral Diseases, Tampere University Hospital. 120 patients who have either recurrent acute or chronic rhinosinusitis without nasal polyposis and whose sinusitis is limited mainly into maxillary sinuses, are recruited in the study. After the first visit, when the patient has filled the consent form and all the preoperative evaluation has been carried out, the examining doctor sends the patient's study number and all the information needed for the randomization and allocation to a person who carries out the randomization and does not know anything else about the patient and does not participate in the examination or the treatment of the patients. The patients are allocated either into the chronic maxillary sinusitis (60 patients) or the recurrent maxillary sinusitis (60 patients) branch of the study. Then, the patients are consecutively randomized into two treatment groups in the proportion of 1 to 1 by using MINIM, an MS-DOS program that randomizes patients to treatment groups by the method of minimization. The treatment groups are A) Balloon sinuplasty group and B) Placebo group (sham surgery).

Sample size calculation was based on comparison of proportions between two independent samples. It was estimated that the balloon sinuplasty could improve the situation of approximately 60% of the chronic rhinosinusitis patients. There is a likely placebo effect in the sham surgery group and therefore it was estimated that the situation in 20% of the patients in that group could significantly be improved. When using alfa = 0.05, power = 0.80 and the proportion difference of 60% vs. 20%, the calculation showed that 27 + 27 observations are needed. This was rounded up to final sample of 30 patients in the balloon sinuplasty group and 30 patients in the placebo group. Similar benefits of balloon sinuplasty were assumed concerning recurrent acute maxillary rhinosinusitis and therefore the final sample size would also be 30 patients in the balloon sinuplasty group and 30 patients in the placebo group. The total sample size will therefore be 120 patients.

The treatment is performed in similar circumstances for both the balloon sinuplasty and the placebo group in the day surgery section of the ENT clinic. The staff of the day surgery section is instructed to avoid any kind of communication, before and during the operation as well as during the post-operative care, which might reveal the group of the patient. The operation theatre nurses open the sealed randomization envelope and prepare the room according to it. All the surgical devices to be used in the operation are hidden under a sterile linen when the patient enters the room. Before the operation begins, the patient is set on the operation table and his/her eyes are covered with moist gauze dressing pads. The operating doctor reads the randomization group status information from the envelope, which tells whether the operation is going to be a balloon sinuplasty or a placebo procedure, in the operation theatre just before the operation.

The operations are carried out in local anesthesia which is always performed similarly for both groups. Topical anesthesia is performed for each patient. All the procedures are performed under a direct vision of a straight, 4mm diameter, 0-degree endoscope. Operation time and possible bleeding and pain during the operation are documented. Nasal mucosal biopsies are taken from the anterior portions of middle turbinates from all the patients. Then in the Balloon sinuplasty group the balloon sinuplasty operation is performed: the shapeable tip of the balloon dilatation device (Entellus XprESS LoProfile; Stryker Corporation, Kalamazoo, Michigan, U.S.A.), with maxillary bending, is inserted into the maxillary sinus ostium. Then guided with the tip, a flexible balloon (6 mm x 20 mm) is gently inserted into the ostium and inflated up to 12 atm for 15 seconds. The dilatation is repeated one more time. The same procedure is performed for both maxillary sinuses. In the placebo treatment group the middle meatus is gently palpated with a curved suction tip (the tip is not connected to a suction unit). The curved suction tip is placed medial to the uncinate process. In order to create a better placebo effect, the operating doctor says: "Now inflate the balloon up to 12 atm for 15 seconds." After 15 seconds the doctor says: "Deflate the balloon." This is repeated one more time. Similar procedure is carried out on both sides.

The operating doctor does not participate in the pre- or postoperative evaluation of the patients. The information, whether the patient had a placebo procedure or the balloon sinuplasty procedure, is not written in the patient's medical record. It is only written that the patient had an operation in accordance with the study protocol. The more detailed information of the operation is written on the Surgery form and the form is sealed in an envelope and the envelope is sent to the study nurse, who stores it inside a locked filing cabinet in her locked office. The envelope is only opened in the end of the 12-month follow-up visit.

The examining doctor follows the patients for the next 12 months after the operation. The follow-up visits take place 3 and 12 months postoperatively. At 6 and 9 months postoperatively, there will be a phone interview by the study nurse and the patients will fill a web based electronic follow-up form. In the end of the 12 month follow-up visit, the examining doctor and the patient are informed about the patient's group status and the patients in the placebo group are given the option to receive the balloon sinuplasty treatment outside the study.

The effect of balloon sinuplasty treatment in chronic maxillary rhinosinusitis will be measured primarily with the Sino-Nasal Outcome Test (SNOT-22), which measures the quality of life and also the outcome of a surgical intervention. In recurrent acute maxillary rhinosinusitis, the effect of balloon sinuplasty treatment will be measured primarily with the number of acute rhinosinusitis infections. Besides this, number of antibiotic treatments and sick leaves are inquired, Visual Analog Scale (VAS) is used, rhinomanometry, nasal endoscopy and general evaluation of the patients clinical ORL-status are performed. Cone Beam Computed Tomography (CBCT) is performed preoperatively and at the 12 month follow-up visit. To measure the Eustachian tube dysfunction, patients are going to fill in the Eustachian Tube Dysfunction Questionnaire (ETDQ-7) and tympanometry and tubomanometry are performed. To estimate the histological effectiveness for rhinal inflammation, pre- and postoperative biopsies are taken from the middle turbinates.

In chronic maxillary rhinosinusitis, the improvement of the quality of life will be analysed with either paired t-test or Wilcoxon rank sum test depending on the shape of the distribution of the SNOT-22 scores. The comparison between the groups regarding the SNOT-22 score change will be carried out with either independent samples T-test or Mann-Whitney test depending on the distribution. In recurrent acute maxillary rhinosinusitis, the reduction of sinusitis episodes and comparison between two groups will be analysed with Fisher exact test.

The results of this study will be submitted for publication to peer reviewed international journals.

The Pirkanmaa Hospital District and the research group with its grants bear the expenses of the study. The researchers are not payed for executing the study but they will apply for grants.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old and younger than 70 years old
* Patients willing to participate in the study
* Patients whose diseases fill the definitions of chronic or acute recurrent maxillary rhinosinusitis
* Patients with chronic maxillary rhinosinusitis has not responded to a 3-month trial of topical corticosteroid treatment
* SNOT-22 points 8 or more in chronic maxillary rhinosinusitis
* In recurrent acute maxillary rhinosinusitis, no SNOT-22 point limits are used
* Modified Lund-Mackay inclusion criteria in chronic rhinosinusitis group:

  1. Maxillar 0-2
  2. Anterior Ethmoid 0-2
  3. Posterior Ethmoid 0-1
  4. Sphenoid 0-1
  5. Frontal 0-1
  6. Ostiomeatal complex 0 or 2

Exclusion Criteria:

* Chronic rhinosinusitis with nasal polyps
* Notable inflammation in the ethmoidal, sphenoidal or frontal sinuses along with maxillary sinusitis
* Previous nasal surgery
* Sinonasal tumor
* Maxillary rhinosinusitis caused by a dental problem
* Facial pain caused by other etiologies
* Cystic fibrosis
* Gross immunodeficiency
* Congenital mucociliary problems
* Non-invasive fungal balls and invasive fungal disease
* Systemic vasculitis and granulomatous disease
* Severe systemic diseases
* Malignancies
* Pregnancy

Definitions:

Recurrent acute maxillary rhinosinusitis:

* 4 or more episodes (< 12 weeks) of acute rhinosinusitis with typical symptoms per year and no persistent symptoms between the rhinosinusitis episodes (Chan and Kuhn 2009)
* The diagnosis of the recurrent episodes of acute rhinosinusitis have been made with the following criteria:

  * Increase of symptoms after 5 days or persistent symptoms after 10 days and
  * During the episode, 2 or more symptoms, one of which should be either nasal blockage/obstruction or nasal discharge (anterior/posterior nasal drip)
  * +/- facial pain/pressure
  * +/- reduction or loss of smell (Fokkens et al. 2012) and either
  * Signs of mucopurulent discharge primarily from the middle meatus seen in anterior rhinoscopy or nasoendoscopy and/or
  * Oedema/mucosal obstruction primarily seen in the middle meatus in anterior rhinoscopy or nasoendoscopy and/or
  * Signs of mucopurulent discharge seen in the nasopharynx or posterior oropharynx and/or
  * Signs of acute maxillary sinusitis is seen in sinus X-rays or CT/CBCT scans and/or
  * Signs of acute maxillary sinusitis seen in the sinus ultrasound
* No signs of mucosal disease at nasoendoscopy during the asymptomatic period
* At most, minor signs of inflammation in the maxillary sinuses and/or ostiomeatal complex in CT/CBCT scans during the asymptomatic period

  * Maximum 2-3 mm mucosal thickness in maxillary sinus medial and lateral wall

Chronic maxillary rhinosinusitis:

* Presence of typical symptoms of chronic rhinosinusitis for equal or longer than 12 weeks

  * 2 or more symptoms, one of which should be either nasal blockage/obstruction or nasal discharge (anterior/posterior nasal drip)
  * +/- facial pain/pressure
  * +/- reduction or loss of smell and either
  * Endoscopic signs of mucopurulent discharge primarily from middle meatus and/or
  * Endoscopic signs of oedema/mucosal obstruction primarily in middle meatus and/or
  * Inflammatory mucosal changes within the ostiomeatal complex and/or sinus in the CT/CBCT scans and the changes are limited mainly into maxillary sinuses (Fokkens et al. 2012)

The patients are not recruited in the study while they are having an exacerbation of chronic rhinosinusitis or an ongoing acute rhinosinusitis. Neither are the follow-up visits carried out during these episodes but postponed later. This way it can be ensured that the preoperative evaluation and the follow-up evaluation correspond with each other.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Sino-Nasal Outcome Test (SNOT-22) score at 3 months | Patients fill the SNOT-22-questionnaire preoperatively and 3 months post-operative
  The effect of balloon sinuplasty treatment in chronic maxillary rhinosinusitis is measured primarily with the Sino-Nasal Outcome Test (SNOT-22). The Sino-Nasal Outcome Test (SNOT-22) is a patient-reported measure of outcome developed for use in chronic rhinosinusitis with or without nasal polyposis. It can be used to assess the impact of chronic rhinosinusitis on the patient's quality of life. It may also be used to measure the outcome of a surgical intervention (Hopkins et al. 2009). In this study, SNOT-22 translated in Finnish is used. The validation of the Finnish version has been made by the Finnish Medical Society Duodecim.
Change from baseline Sino-Nasal Outcome Test (SNOT-22) score at 6 months | Patients fill the SNOT-22-questionnaire preoperatively and 6 months post-operative
  The effect of balloon sinuplasty treatment in chronic maxillary rhinosinusitis is measured primarily with the Sino-Nasal Outcome Test (SNOT-22). The Sino-Nasal Outcome Test (SNOT-22) is a patient-reported measure of outcome developed for use in chronic rhinosinusitis with or without nasal polyposis. It can be used to assess the impact of chronic rhinosinusitis on the patient's quality of life. It may also be used to measure the outcome of a surgical intervention (Hopkins et al. 2009). In this study, SNOT-22 translated in Finnish is used. The validation of the Finnish version has been made by the Finnish Medical Society Duodecim.
Change from baseline Sino-Nasal Outcome Test (SNOT-22) score at 9 months | Patients fill the SNOT-22-questionnaire preoperatively and 9 months post-operative
  The effect of balloon sinuplasty treatment in chronic maxillary rhinosinusitis is measured primarily with the Sino-Nasal Outcome Test (SNOT-22). The Sino-Nasal Outcome Test (SNOT-22) is a patient-reported measure of outcome developed for use in chronic rhinosinusitis with or without nasal polyposis. It can be used to assess the impact of chronic rhinosinusitis on the patient's quality of life. It may also be used to measure the outcome of a surgical intervention (Hopkins et al. 2009). In this study, SNOT-22 translated in Finnish is used. The validation of the Finnish version has been made by the Finnish Medical Society Duodecim.
Change from baseline Sino-Nasal Outcome Test (SNOT-22) score at 12 months | Patients fill the SNOT-22-questionnaire preoperatively and 12 months post-operative
  The effect of balloon sinuplasty treatment in chronic maxillary rhinosinusitis is measured primarily with the Sino-Nasal Outcome Test (SNOT-22). The Sino-Nasal Outcome Test (SNOT-22) is a patient-reported measure of outcome developed for use in chronic rhinosinusitis with or without nasal polyposis. It can be used to assess the impact of chronic rhinosinusitis on the patient's quality of life. It may also be used to measure the outcome of a surgical intervention (Hopkins et al. 2009). In this study, SNOT-22 translated in Finnish is used. The validation of the Finnish version has been made by the Finnish Medical Society Duodecim.
Change from baseline in the number of acute rhinosinusitis infections at 3 months | Preoperative and 3 months post-operative
  In recurrent acute maxillary rhinosinusitis, the effect of balloon sinuplasty treatment is measured primarily with the change in number of acute rhinosinusitis infections. It is hard to measure the effect of the balloon sinuplasty in recurrent acute rhinosinusitis with methods questioning the current state of disease, because patients are asymptomatic between episodes of sinusitis. That is why the patients are asked the number of maxillary rhinosinusitis during the last 3 months preoperatively and that number is compared to the number of postoperative maxillary rhinosinusitis asked at 3 months after the operation.
Change from baseline in the number of acute rhinosinusitis infections at 6 months | Preoperative and 6 months post-operative
  In recurrent acute maxillary rhinosinusitis, the effect of balloon sinuplasty treatment is measured primarily with the change in number of acute rhinosinusitis infections. It is hard to measure the effect of the balloon sinuplasty in recurrent acute rhinosinusitis with methods questioning the current state of disease, because patients are asymptomatic between episodes of sinusitis.
  The patients are asked the number of maxillary rhinosinusitis during the last 6 months preoperatively and that number is compared to the number of postoperative maxillary rhinosinusitis that the patients have had during the post-operative 6 months.
Change from baseline in the number of acute rhinosinusitis infections at 12 months | Preoperative and 12 months post-operative
  In recurrent acute maxillary rhinosinusitis, the effect of balloon sinuplasty treatment is measured primarily with the change in number of acute rhinosinusitis infections. It is hard to measure the effect of the balloon sinuplasty in recurrent acute rhinosinusitis with methods questioning the current state of disease, because patients are asymptomatic between episodes of sinusitis.
  The patients are asked the number of maxillary rhinosinusitis during the last 12 months preoperatively and that number is compared to the number of postoperative maxillary rhinosinusitis infections that the patients have had during the post-operative 12 months.

SECONDARY OUTCOMES:
Amount of sick leaves | Preoperative and 3, 6, 9 and 12 months post-operative
  The number of sick leaves during the last year, last 6 and last 3 months is asked preoperatively, focusing on the sick leaves that are caused because of chronic or recurrent rhinosinusitis. Also, the information about the postoperative sick leaves is collected during all the controls in order to find out whether the amount of sick leaves changes after the operation or not.
Number of antibiotic treatments needed | Preoperative and 3, 6, 9 and 12 months post-operative
  One way to estimate the effectiveness of balloon sinuplasty is to collect the data of antibiotic treatments. Especially in the cases of recurrent acute rhinosinusitis this is valid information. In this study, the number of antibiotic treatments during the last year, last 6 and last 3 months is checked from the Prescription Centre. Also, the information about the postoperative antibiotic treatments is collected during all the controls from the Prescription Centre in order to find out whether the amount of antibiotic treatments changes after the operation or not.
Eustachian Tube Dysfunction Questionnaire (ETDQ-7) | Preoperative and 3, 6, 9 and 12 months post-operative
  Eustachian tube dysfunction is a common condition which causes ear symptoms such as clogging and popping. The condition is also commonly associated with chronic sinusitis. The ETDQ-7 is a valid and reliable symptom score for use in adult patients with Eustachian tube dysfunction. It is a 7-item questionnaire which inquires patient´s ear symptoms. It is easily administered in the clinical setting and has minimal burden to respondents (McCoul et al. 2012). In this study ETDQ-7 is used to evaluate patient´s possible ear symptoms which refer to Eustachian tube dysfunction. Patients fill the ETDQ-7-questionnaire preoperatively and during all the controls.
Visual Analog Scale (VAS) | Preoperative and 3, 6, 9 and 12 months post-operative
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left-hand end of the line to the point that the patient marks (Wewers and Lowe 1990). In this study, VAS is used to measure the symptoms of nasal obstruction, nasal discharge, facial pain/pressure and olfactory disorder. Patients report their symptoms preoperatively and during all the controls.
The clinical status of nasal mucosa in nasal endoscopy assessed in terms of mucosal oedema, nasal discharge and synechiae | Preoperative and during post-operative visits at 3 and 12 months
  Nasal endoscopy involves evaluation of the nasal and sinus passages with direct vision. It is a commonly performed procedure in the otolaryngology and serves as an objective diagnostic tool in the evaluation of nasal mucosa, sinonasal anatomy, and nasal pathology. During the diagnostic nasal endoscopy, a patient is always awake and seated upright in a chair. A local anaesthetic lidocaine spray is applied to the nose to make insertion of the endoscope less uncomfortable. In this study, nasal endoscopy is done to assess nasal mucosa preoperatively and during postoperative visits at 3 and 12 months. Mucosal oedema, nasal discharge and synechiae are documented and reported either "Yes" or "No". A special attention is paid on the findings in the middle meatus of the nose.
Signs of Eustachian tube dysfunction in otomicroscopic ear status | Preoperative and during post-operative visits at 3 and 12 months
  In clinical examination, preoperatively and during the control visits at 3 and 12 months, a special attention is paid on the otomicroscopic ear status in order to find out signs of Eustachian tube dysfunction, such as tympanic membrane retraction and middle ear effusion. The tympanic membrane retraction and the presence of middle ear effusion are categorized either "Yes" or "No" and evaluated for both ears separately. Valsalva and Toynbee tests are also performed during the examination and documented either "positive" or "negative" for both ears separately.
Inspiratory nasal resistance in Rhinomanometry | Preoperative and during post-operative visits at 3 and 12 months
  Rhinomanometry measures the nasal airway resistance and flow. It is a tool for determining the degree of airflow obstruction before and after surgical procedures and medical interventions. It may also help to distinguish functional causes of upper airway obstruction from structural causes (Clement et al. 2014). Active anterior rhinometry is the most commonly used method and it is performed as follows: One nostril is closed with an adhesive tape, pierced by the catheter for pressure determination, and a mask covers the nose and the mouth. The pressure flow curve is recorded with a storage oscilloscope and projected onto a pre-printed diagram. In this study, the rhinomanometry is used to evaluate the possible effect of balloon sinuplasty procedure on the nasal airway resistance. The total inspiratory nasal resistance is measured as well as the resistance in right and left nostrils separately. The measurement is carried out preoperatively and during the control visits at 3 and 12 months.
Signs of Eustachian tube dysfunction in Tympanometry | Preoperative and during post-operative visits at 3 and 12 months
  In tympanometry, middle ear pressure is measured with an electroacoustic impedance meter that allows the precise evaluation of eardrum mobility and helps to assess Eustachian tube function. The tympanometric curves are traditionally classified as follows (Lidén 1969; Jerger 1970): type A, normal ET function; type B, flat tympanogram characteristic of the presence of fluid in the middle ear or eardrum perforation; or type C, peak at very negative pressure, typically 150 dPa, which may be indicative of eardrum retraction and Eustachian tube dysfunction. Tympanometric peak pressure is the peak admittance in the tympanogram and an indirect measurement of middle ear pressure. In this study, the tympanometric peak pressure is measured and the type of tympanometric curve is recorded from both ears separately. The measurement is carried out preoperatively and during the control visits at 3 and 12 months.
The opening of Eustachian tube in Tubomanometry | Preoperative and during post-operative visits at 3 and 12 months
  The principle of tubomanometry is to deliver defined pressures of 30, 40 and 50 mbar to the epipharynx through a nasal applicator. If the Eustachian tube opens during swallowing, the defined pressure applied to the epipharynx is transmitted to the middle ear and the pressure change can be registered in the external auditory canal. In this study the opening latency index (R-value) is recorded in pressures of 30, 40 and 50 mbar for both ears separately and also the information, whether the Eustachian tube opened or not in those pressures. The opening latency index (R-value) reflects the latency between pressure application in the epipharynx and measurement of a pressure change in the ear canal. An immediate opening (R < 1) indicates normal ET function and a late opening (R ≥ 1) indicates restricted ET function. No opening (R negative or not measurable) indicates complete obstruction of the ET (Schröder et al. 2015).
Change from baseline in Lund-Mackay score at 12 months measured from the Cone Beam Computed Tomography (CBCT) scans | Preoperative and 12 months post-operative
  Cone Beam Computed Tomography (CBCT) is an X-ray based volume acquisition method providing 3D images of the head. In this study CBCT is used preoperatively in the diagnostics of chronic rhinosinusitis in patient selection. Another CBCT scan is taken during the control visit at 12 months.
  The radiological staging (Lund-Mackay score) of the chronic sinusitis is graded from the CBCT scans both preoperatively and postoperatively. When evaluating a CBCT scan of the paranasal sinuses and ostiomeatal complex, the researcher assigns each sinus a score of: 0 (no abnormality), 1 (partial opacification) or 2 (complete opacification).The ostiomeatal complex is assigned a score of either 0 (not obstructed) or 2 (obstructed). Each side is graded separately. A combined score of up to 24 is possible.
Volumetric measurements with OnDemand3D™ software analyzed from Cone Beam Computed Tomography (CBCT) scans | Preoperative and 12 months post-operative
  Cone Beam Computed Tomography (CBCT) is an X-ray based volume acquisition method providing 3D images of the head. In this study CBCT is used preoperatively in the diagnostics of chronic rhinosinusitis in patient selection. Another CBCT scan is taken during the control visit at 12 months.
  Volumetric measurements of the sinuses, infundibuli and ostia will be made from the scans both preoperatively and postoperatively. Volumetric measurements are performed with OnDemand3D™ software (version 1.0, CyberMed, Inc., Yuseong-gu, Daejeon, South Korea) which has been used for similar purpose in a previous study (Valtonen et al. 2018). In accordance with the previous study, the same Hounsfield Unit (HU) values from -1000 to -430 in CBCT scans are utilized to define air in nose for volumetric measurements.
Nasal mucosal biopsy | In the operation and 12 months post-operative
  Nasal mucosal biopsy is taken from the anterior head of both middle turbinates in local anaesthesia in the beginning of the operations and during the post-operative visit at 12 months. In local anaesthesia a local anaesthetic (Lidocain 10mg/ml c. adrenalin, Orion, Finland) is applied to the anterior head of the middle turbinate. All the specimens are examined by a pathologist. The main purpose of the examination is to compare preoperative and post-operative mucosal specimens and evaluate the effect of balloon sinuplasty treatment on the degree of inflammation in the nasal cavity.

OTHER OUTCOMES:
Adverse events | 3, 6, 9 and 12 months post-operative
  Information about possible postoperative adverse events is asked and determined during the clinical post-operative visits at 3 and 12 months. The patients are asked about possible postoperative adverse events also in the web based electronic question forms which the patients fill at 6 and 9 months post-operative.
General evaluation of the patient and clinical ORL-status | Preoperative and during post-operative visits at 3 and 12 months
  Careful ORL-status is made preoperatively and during the postoperative visits at 3 and 12 months. Focus is on the nasal status and especially on the structure, abnormalities and other findings. Careful ear status is also performed because of the interest on the correlation between chronic rhinosinusitis and Eustachian tube dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Rautiainen, Professor, Study Chair — Professor; Johanna Luukkanen, MD, Principal Investigator — Doctoral thesis researcher
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan Y, Kuhn FA. An update on the classifications, diagnosis, and treatment of rhinosinusitis. Curr Opin Otolaryngol Head Neck Surg. 2009 Jun;17(3):204-8. doi: 10.1097/MOO.0b013e32832ac393. PMID 19346944
- [Background] Clement PA, Halewyck S, Gordts F, Michel O. Critical evaluation of different objective techniques of nasal airway assessment: a clinical review. Eur Arch Otorhinolaryngol. 2014 Oct;271(10):2617-25. doi: 10.1007/s00405-013-2870-9. Epub 2014 Jan 20. PMID 24442716
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl. 2012 Mar;23:3 p preceding table of contents, 1-298. PMID 22764607
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Jerger J. Clinical experience with impedance audiometry. Arch Otolaryngol. 1970 Oct;92(4):311-24. doi: 10.1001/archotol.1970.04310040005002. No abstract available. PMID 5455571
- [Background] Liden G. The scope and application of current audiometric tests. J Laryngol Otol. 1969 Jun;83(6):507-20. doi: 10.1017/s0022215100070651. No abstract available. PMID 5785649
- [Background] McCoul ED, Anand VK, Christos PJ. Validating the clinical assessment of eustachian tube dysfunction: The Eustachian Tube Dysfunction Questionnaire (ETDQ-7). Laryngoscope. 2012 May;122(5):1137-41. doi: 10.1002/lary.23223. Epub 2012 Feb 28. PMID 22374681
- [Background] Schroder S, Lehmann M, Korbmacher D, Sauzet O, Sudhoff H, Ebmeyer J. Evaluation of tubomanometry as a routine diagnostic tool for chronic obstructive Eustachian tube dysfunction. Clin Otolaryngol. 2015 Dec;40(6):691-7. doi: 10.1111/coa.12451. PMID 25925071
- [Background] Valtonen O, Bizaki A, Kivekas I, Rautiainen M. Three-Dimensional Volumetric Evaluation of the Maxillary Sinuses in Chronic Rhinosinusitis Surgery. Ann Otol Rhinol Laryngol. 2018 Dec;127(12):931-936. doi: 10.1177/0003489418801386. Epub 2018 Sep 22. PMID 30244583
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679